CLINICAL TRIAL: NCT03822130
Title: A Randomized Controlled Trial for Intra-arterial Infusion Chemotherapy Combined With Sodium Bicarbonate and Systemic Chemotherapy for Unresectable Gastric Cancer
Brief Title: Intra-arterial Infusion Chemotherapy Combined With Sodium Bicarbonate for Unresectable Gastric Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR2018001142
Record Dates: First submitted 2019-01-23; First posted 2019-01-30 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-01

CONDITIONS: Successful Conversion Rate of Operation; Unresectable Gastric Cancer
MeSH Terms: interventions — Sodium Bicarbonate; Neoadjuvant Therapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Placebo Comparator): Systemic Chemotherapy + Oral Chemotherapy Group
  Interventions: Drug: Systemic Chemotherapy; Drug: Oral Chemotherapy
- Group 2 (Experimental): Arterial catheter infusion chemotherapy plus oral chemotherapy group
  Interventions: Drug: Arterial catheter infusion chemotherapy; Drug: Oral Chemotherapy
- Group 3 (Experimental): Arterial catheter infusion chemotherapy + sodium bicarbonate plus oral chemotherapy group
  Interventions: Drug: Arterial catheter infusion chemotherapy; Drug: Sodium Bicarbonate; Drug: Oral Chemotherapy

INTERVENTIONS:
Drug: Arterial catheter infusion chemotherapy — Arterial catheter infusion chemotherapy
  Arms: Group 2; Group 3
Drug: Sodium Bicarbonate — Arterial catheter infusion Sodium Bicarbonate
  Arms: Group 3
Drug: Systemic Chemotherapy — Systemic Chemotherapy
  Arms: Group 1
Drug: Oral Chemotherapy — Oral Chemotherapy

SUMMARY:
This project intends to compare the clinical effects and side effects of three kinds of treatment methods in the treatment of unresectable gastric cancer by intra-arterial catheter infusion chemotherapy combined with sodium bicarbonate and systemic chemotherapy. It is clear that intra-arterial catheter infusion chemotherapy combined with sodium bicarbonate is not suitable for the treatment of unresectable gastric cancer. The clinical practice value of resection of gastric cancer can provide high quality evidence-based medical basis for the treatment guidelines of advanced gastric cancer, and explore a new clinical technology with exact curative effect and higher safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 75 years;
2. Ultrasound gastroscopy or imaging (CT) can diagnose potentially unresectable gastric cancer (T4a-bN2-3M0) with indications of neoadjuvant chemotherapy or transformation therapy;
3. Pathological diagnosis of gastric cancer;
4. No contraindication of chemotherapy;
5. Patients who did not undergo chemotherapy or were diagnosed for the first time.

Exclusion Criteria:

1. Those who fail to comply with the requirements of the trial, obviously violate this regimen, or change to other regimens in the course of treatment;
2. The life expectancy of patients with extensive systemic metastasis is less than 3 months;
3. Leukocyte count is less than 2*109/L and platelet count is less than 75*10^9/L;
4. Severe heart, liver and kidney diseases, unable to tolerate chemotherapy;
5. Patients without gastric cancer complications such as massive gastrointestinal bleeding and perforation need to be treated in emergency department;
6. Patients with distant metastasis (excluding group 16 lymph node metastasis);
7. Patients with other tumors, with a history of malignant tumors (excluding early primary cancers);
8. The patient himself asked to withdraw from the trial;
9. Researchers believe that patients are not suitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful conversion rate of operation | 42 days

SECONDARY OUTCOMES:
ORR | 42 days
  Objective Response rate
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- The Second affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China